CLINICAL TRIAL: NCT04408495
Title: Effect of IntraoperatiVe High Positive End-ExpirAtory Pressure (PEEP) With ReCruitment MAneuveRs vs Low PEEP on Major Postoperative Pulmonary Complications and Death After On-pump Cardiac Surgery in High-risk Patients: the VACARM Study
Brief Title: Intraoperative Mechanical Ventilation and Postoperative Pulmonary Complications After On-pump Cardiac Surgery in High-risk Patients
Acronym: VACARM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC18_8854_VACARM
Record Dates: First submitted 2020-05-15; First posted 2020-05-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pulmonary Complications
Keywords: recruitment maneuvers; Postoperative pulmonary complications; Peep; Cardiac surgery; Mortality
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, comparative, parallel-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group_MRA (Experimental): Recruitment maneuvers and high PEEP
  Interventions: Procedure: Intervention group_MRA
- Control group (Active Comparator): No recruitment maneuvers and low PEEP
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Intervention group_MRA — Tidal Volume (Vt) =6-8 mL/kg of predicted body weight (PBW), Peep=8 cmH2O, recruitment maneuvers=30cm H2O every 30 min after intubation (except during CPB), after any disconnection and at the admission in ICU.
  Recruitment maneuvers are performed in accordance with the surgical team an if SAP≥90 mmHg or MAP≥65 mmHg.
  Ventilation is maintained during CPB Vt=2.5 mL/kg, Peep= 5 cmH2O
  Other Names: recruitment maneuvers
  Arms: Intervention group_MRA
Procedure: Control group — Vt=6-8 mL/kg of PBW, Peep=5 cmH2O , No recruitment maneuvers. Ventilation maintained during CPB Vt=2.5 mL/kg, Peep= 5 cmH2O.
  Other Names: NO recruitment maneuvers
  Arms: Control group

SUMMARY:
Controversies remain concerning the best intraoperative mechanical ventilation regimen for major cardiac surgery. While the use of intra operative low tidal volumes is now standard practice, the optimal level of positive end-expiratory pressure (PEEP) and the use of recruitment maneuvers (RM) remain controversial. The aim of this study is to compare two regimens of intraoperative mechanical ventilation on postoperative outcomes in cardiac surgery patients at risk of postoperative pulmonary complications

DETAILED DESCRIPTION:
In this randomized controlled trial, cardiac surgery patients at risk of postoperative pulmonary complications will be assigned to intraoperative ventilation with high PEEP and RM or intraoperative mechanical ventilation with low PEEP and without RM. The primary endpoint will be a composite endpoint including major postoperative complications within the first postoperative week and death within the 28 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years-old,
* Evaluated before cardiopulmonary bypass for any cardiac surgical procedure (e.g. coronary artery bypass grafting, valve, aorta, or combined procedures),
* With a pulmonary risk score ≥ 2
* Who gave written informed consent
* affiliated to a social security system

Exclusion Criteria:

* BMI > 40kg/m2 ;
* Left Ventricular Ejection Fraction < 35% ;
* Preoperative shock ;
* Aortic surgery with planned circulatory arrest ;
* Minimally invasive cardiac surgery ;
* Emergency surgery with patient unable to give written informed consent
* Heart transplantation
* Mechanical circulatory support surgery
* Pregnant or lactating women
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of major pulmonary complications and death | 28 days after surgery
  Major pulmonary complications, defined as prolonged mechanical ventilation >24h post-operatively, pneumonia (defined according to the 2017 French guidelines) or reintubation for any cause within 7 post-operative days, or death

SECONDARY OUTCOMES:
Rate of patients with hypotension | intraoperative period
  Safety criteria with Hypotension lasting more than 60 seconds after the end of the recruitment maneuvers
Evaluate the postoperative blood gases | 30 minutes after extubation
  Measure of PaO2 (mmHg)
Evaluate the postoperative blood gases | 30 minutes after extubation
  Measure of HCO3 (mmol/l)
Evaluate the postoperative blood gases | 30 minutes after extubation
  Measure of PaCO2 (mmHg)
Evaluate the postoperative blood gases | 30 minutes after extubation
  Measure of SaO2 (%)
Evaluate the postoperative blood gases | Day 1
  Measure of PaO2 (mmHg)
Evaluate the postoperative blood gases | Day 1
  Measure of HCO3 (mmol/l)
Evaluate the postoperative blood gases | Day 1
  Measure of PaCO2 (mmHg)
Evaluate the postoperative blood gases | Day 1
  Measure of SaO2 (%)
Evaluate the postoperative blood gases | Day 2
  Measure of PaO2 (mmHg)
Evaluate the postoperative blood gases | Day 2
  Measure of HCO3 (mmol/l)
Evaluate the postoperative blood gases | Day 2
  Measure of PaCO2 (mmHg)
Evaluate the postoperative blood gases | Day 2
  Measure of SaO2 (%)
Pulmonary function tests | Day -1 or Day 0
  Measure of vital capacity (CV) and maximum expiratory volume by second (VEMS) by spirometry
Pulmonary function tests | Day 3
  Measure of vital capacity (CV) and maximum expiratory volume by second (VEMS) by spirometry
Pulmonary function tests | Day 5
  Measure of vital capacity (CV) and maximum expiratory volume by second (VEMS) by spirometry
Daily evaluation of organ failure | Up to 7 days
  SOFA score
Daily evaluation of delirium | Up to 7 days
  CAM-ICU scale
Rate of Postoperative pulmonary complications (PPC) | within the 28 days after surgery
  Pneumonia (defined according to the 2017 French guidelines), re-intubation within 7 days, mechanical ventilation >24h, pneumothorax, Atelectasis, Acute Respiratory Distress Syndrome. PPC grade (according to Huzelbos et al; JAMA)
Rate of Postoperative non pulmonary complications | within the 28 days after surgery
  Re intervention for acute bleeding, Pericardial Tamponade, Sternal wound infection, Ventricular Arrhythmia, Atrial fibrillation, Myocardial infarction, Mesenteric ischemia, Sepsis/septic shock, Acute kidney injury with renal replacement therapy
Ventilation duration, length of stay in ICU and in the study hospital and death | Day 28
  Number of Ventilatory-free days, vasopressor-free days, Renal Replacement Therapy free days, ICU-free days and hospital-free days
Mortality rate | Day 28
Mortality rate | Day 90
Mortality rate | Day 180
Biomarkers of systemic inflammation and of epithelial and endothelial aggression | Day 0
  Plasma levels of TNFα, IL1β, IL6, IL8 et IL10, Angiopoeitin 2 and soluble form of receptor for advanced glycation end products (sRAGE)
Biomarkers of systemic inflammation and of epithelial and endothelial aggression | Day 1
  Plasma levels of TNFα, IL1β, IL6, IL8 et IL10, Angiopoeitin 2 and soluble form of receptor for advanced glycation end products (sRAGE)
Length of stay in ICU and in the study hospital | Day 180
  Number of days in ICU and in the study hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie DEMAURE, Principal Investigator — CHU Rennes; Nicolas NESSELER, MD, Principal Investigator — CHU Rennes
Locations (10):
- France (10):
  - CHU Amiens-Picardie, Amiens
  - CHRU Brest, Brest
  - CHU de Dijon, Dijon
  - CHU de Nancy, Nancy
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU Nantes, Saint-Herblain
  - CHU de Toulouse, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after the primary publication of the results, to any researchers who provide a methodologically sound proposal. Proposals should be directed to dri@chu-rennes.fr. To gain access, data requestors will need to sign a data access agreement; depending on the case, additional formalities may be required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data availability after the primary publication of the results and until the database is deleted
Access Criteria: Any researchers who provide a methodologically sound proposal will be able to access the IPD ans supporting information. To gain access, data requestors will need to sign a data access agreement; depending on the case, additional formalities may be required.

REFERENCES:
- [Derived] Demaure N, Le Cunff J, Duchene M, Rozec B, Espitalier F, Cabon JM, Oilleau JF, Guerci P, Labaste F, Abou-Arab O, Guinot PG, Duval P, Besnier E, Flecher E, Leroyer I, Morcet J, Fougerou-Leurent C, Mansour A, Nesseler N; VACARM investigators; ATLANREA study group. Impact of intraoperatiVe moderAte positive end-expiratory pressure with reCruitment mAnoeuvres versus low positive end-expiRatory pressure on major postoperative pulMonary complications and death after on-pump cardiac surgery in high-risk patients: the VACARM randomised clinical trial-study protocol. BMJ Open. 2025 Oct 29;15(10):e104179. doi: 10.1136/bmjopen-2025-104179. PMID 41161829